CLINICAL TRIAL: NCT00134927
Title: Usage Patterns of OTC Nicotine Patches: Consumer Survey
Brief Title: A Survey on Consumer Use of Over-the-Counter (OTC) Nicotine Patches
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Chih-Wen Shi, MD, University California, San Diego
Other Study IDs: NIDA-15853-1; K23-15853-1; DPMC
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2008-10

CONDITIONS: Nicotine Dependence; Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Since 1996, the nicotine patch has been re-classified from prescription to over-the-counter (OTC) status in the United States. Little is known about how the public uses the OTC nicotine patch due to lack of monitoring. The purpose of this observational study is to describe the characteristics of consumers who purchase OTC nicotine patches from community pharmacies and to determine the factors associated with the appropriate use of nicotine patches.

DETAILED DESCRIPTION:
The nicotine patch is an effective aid for smoking cessation. Since 1996, the nicotine patch has been re-classified from prescription to over-the-counter (OTC) status in the United States. Unlike prescription medications, post-marketing surveillance does not exist for OTC medications. The purpose of this study is to describe the characteristics of consumers who purchase OTC nicotine patches from community pharmacies and to determine the factors associated with appropriate use of nicotine patches.

This prospective, cross-sectional, observational study will include a survey of 600 consumers who purchase OTC nicotine patches at a random sample of 30 community retail pharmacies. Consumers will be recruited by an ad located in the pharmacy next to the nicotine patch product. Participants will fill out a self-administered, anonymous questionnaire at the time of OTC nicotine patch purchase at the pharmacy counter. The questionnaire will gather information about demographics, medical history, smoking history, attitudes toward the nicotine patch, and motivation to quit smoking. No study visits will be required for this study.

ELIGIBILITY:
Inclusion Criteria:

* Purchased OTC nicotine patch (NicoDerm CQ Step I, II, III or Sav-on Nicotine Patch) for personal use

Exclusion Criteria:

* Purchased OTC nicotine patch for someone other than self (e.g., friend or family member)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 600 consumers who purchased over-the-counter nicotine patches from a random sample of 30 retail pharmacies in San Diego County
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2005-09; Primary Completion 2006-05 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Wen Shi, M.D., M.S., Principal Investigator — University of California, San Diego
Locations (1):
- Department of Family and Preventive Medicine, La Jolla, California, United States